CLINICAL TRIAL: NCT05421819
Title: Design and Development of a Novel Food Supplement for Osteoporosis Based on Gut Microbiome Mechanisms: Efficacy and Tolerability Assessment
Brief Title: Design and Development of a Novel Food Supplement for Osteoporosis Based on Gut Microbiome Mechanisms
Acronym: OSTEOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: National Hellenic Research Foundation (Other)
Responsible Party: Principal Investigator, EFSTATHIOS CHRONOPOULOS, Associate Professor in Orthopaedics at National and Kapodistrian University of Athens, Laboratory for Research of the Musculoskeletal System Director, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3847/22.03.2022
Record Dates: First submitted 2022-05-26; First posted 2022-06-16 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Osteopenia; Postmenopausal Osteopenia
Keywords: Dietary supplement for osteopenia; Calcium and vitamin D supplement; Calcium, vitamin D and prebiotics supplement; Calcium, vitamin D, prebiotics and flavonoids supplement; Bone turnover markers; Bone mineral density; Volumetric bone mineral density; Bone geometry; Postmenopausal osteopenia; Gut microbiota analysis
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Calcium and vitamin D supplement (Active Comparator): In this arm, 50 women will receive calcium and vitamin D supplement once per day.
  Interventions: Dietary Supplement: Calcium and vitamin D supplement
- Calcium, vitamin D and prebiotic supplement (Active Comparator): In this arm, 50 women will receive calcium, vitamin D and prebiotic supplement once per day.
  Interventions: Dietary Supplement: Calcium, vitamin D and prebiotic supplement
- Calcium, vitamin D, prebiotic and flavonoid supplement (Active Comparator): In this arm, 50 women will receive calcium, vitamin D, prebiotic and flavonoid supplement once per day.
  Interventions: Dietary Supplement: Calcium, vitamin D and flavonoid supplement

INTERVENTIONS:
Dietary Supplement: Calcium and vitamin D supplement — One hundred fifty postmenopausal women with osteopenia will be randomly and blindly allocated to receive in of the 3 different dietary supplements once per day. Patients of group A will receive orally 600 mg calcium and 2400 IU vitamin D3, group B will receive the same dose of calcium and vitamin D3 plus prebiotics once per day and group C will receive the same dose of calcium, vitamin D3 plus flavonoids once per day.
  Arms: Calcium and vitamin D supplement
Dietary Supplement: Calcium, vitamin D and prebiotic supplement — One hundred fifty postmenopausal women with osteopenia will be randomly and blindly allocated to receive in of the 3 different dietary supplements once per day. Patients of group A will receive orally 600 mg calcium and 2400 IU vitamin D3, group B will receive the same dose of calcium and vitamin D3 plus prebiotics once per day and group C will receive the same dose of calcium, vitamin D3 and flavonoids once per day.
  Arms: Calcium, vitamin D and prebiotic supplement
Dietary Supplement: Calcium, vitamin D and flavonoid supplement — One hundred fifty postmenopausal women with osteopenia will be randomly and blindly allocated to receive in of the 3 different dietary supplements once per day. Patients of group A will receive orally 600 mg calcium and 2400 IU vitamin D3, group B will receive the same dose of calcium and vitamin D3 plus prebiotics once per day and group C will receive the same dose of calcium, vitamin D3 and flavonoids once per day.
  Arms: Calcium, vitamin D, prebiotic and flavonoid supplement

SUMMARY:
It is well proven that the intestinal microbe regulates bone metabolism by the absorption of calcium and other metallic trace elements. Studies also show that regulation of the intestine and its microbe can affect bone density and resistance to a variety of animal models and humans. At the same time, interest in polyphenol-intestinal microbial interactions and in particular flavonoids and catechins has increased. Indeed, it has been observed that they are transformed via the microbe into bioactive compounds, and polyphenols themselves can modify the synthesis of the intestinal microbe.

OSTEOME aspires to design and develop a novel dietary supplement for osteoporosis, activating the intestinal microbiome. At the same time companion biomarkers will be studied related to the efficacy and tolerability of the new supplement. The selection of flavonoids will take place through in vitro and in silico studies focusing on their interaction with pathways that regulate the activity of osteoclasts and osteoblasts. The efficacy and tolerability of the dietary supplement will be evaluated through a randomized clinical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* T-score in the osteopenic range (-1.0 > T-score > -2.5) at either the lumbar spine (LS) or femur as measured by dual energy X-ray absorptiometry (DXA)

Exclusion Criteria:

* T-score in the osteoporotic range (T-score < -2.5) at any site
* Patients receiving supplements of calcium and/or vitamin D at that time or during the last 6 months
* Patients receiving medications known to positively or negatively affect bone turnover or BMD at that time or during the last 3 years (e.g. antiresorptive agents, oestrogens, systemic corticosteroids), or
* Secondary cause of osteoporosis (e.g. alcohol abuse, thyrotoxicosis etc)
* Patients who did not attend to their follow-up appointment and consequently had only the baseline measurements

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women with osteopenia
Enrollment: 117 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Bone geometry | 0 to 12 months
  The primary endpoint is the within and between group change of bone geometry after 12 months of supplementation assessed by peripheral quantitative computed tomography (pQCT) of the tibia

SECONDARY OUTCOMES:
Areal bone mineral density (aBMD), trabecular bone score (TBS), adverse effects (tolerability) and adherence to dietary supplement after 12 months | 12 months
  The secondary endpoints is the within- and between-groups differences of the areal BMD (aBMD) at the lumbar spine (LS) and the total hip (TH) using dual-energy X-ray absorptiometry (DXA) and trabecular bone score (TBS) at LS, and the between-group comparison of the adverse effects (tolerability) and adherence to dietary supplement after 12 months.
Bone turnover markers, PINP and CTX | 3, 6 and 12 months
  Secondary endpoint is the within- and between-group comparison change of bone turnover markers after 3, 6 and 12 months of supplementation.
Change of serum TNF-α, IL-1, OPG, RANKL and IGF-1 | 3, 6 and 12 months
  Secondary endpoint is the within- and between-group comparison change of TNF-α, IL-1, OPG, RANKL and IGF-1 after 3, 6 and 12 months of supplementation.
Change of microMR1 Change of serum miRNAs | 3, 6 and 12 months
  Secondary endpoint is the within- and between-group comparison change of miRNAs after 3, 6 and 12 months of supplementation.
Change of gut microbiota | 12 months
  Secondary endpoint is the within- and between-group comparison change of gut microbiota after 12 months of supplementation.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory for Research of the Musculoskeletal System, Kifissia, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided